CLINICAL TRIAL: NCT00000142
Title: Studies of the Ocular Complications of AIDS (SOCA)--HPMPC Peripheral CMV Retinitis Trial (HPCRT)
Acronym: HPCRT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Baylor College of Medicine (Other); Johns Hopkins University (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Icahn School of Medicine at Mount Sinai (Other); New Jersey Medical School (Other); NYU Langone Health (Other); Northwestern University (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of Miami (Other); University of North Carolina, Chapel Hill (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-41
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Results first posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections; CMV Cytomegalovirus Retinitis
MeSH Terms: conditions — HIV Infections; Cytomegalovirus Retinitis | interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- treatment deferral (Experimental): IV (in the vein) treatment deferred until retinitis progressed, either:
  5 mg/kg IV (in the vein) of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks, or
  5mg/kg IV (in the vein) once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
  Interventions: Drug: Cidofovir
- Cidofovir (low dose) (Experimental): 5 mg/kg IV (in the vein) of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks
  Interventions: Drug: Cidofovir
- Cidofovir (high dose) (Experimental): 5mg/kg IV (in the vein) once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
  Interventions: Drug: Cidofovir

INTERVENTIONS:
Drug: Cidofovir — Three groups:
  1. the deferral group, treatment deferred until retinitis progressed
  2. Low-dose cidofovir group, 5 mg/kg of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks.
  3. High-dose cidofovir group, 5mg/kg once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
  Other Names: Vistide

SUMMARY:
To test and evaluate the efficacy and safety of intravenous cidofovir (Vistide, previously known as HPMPC) for the treatment of retinitis.

DETAILED DESCRIPTION:
CMV (cytomegalovirus) retinitis is the most common intraocular infection in patients with AIDS and is estimated to affect 35 percent to 40 percent of patients with AIDS. Untreated CMV (cytomegalovirus) retinitis is a progressive disorder, the end result of which is total retinal destruction and blindness. As of September 1997, drugs approved by the United States Food and Drug Administration (FDA) for the treatment of CMV (cytomegalovirus)retinitis were ganciclovir (Cytovene), foscarnet (Foscavir), and cidofovir (Vistide). Cidofovir has a prolonged duration of effect permitting intermittent administration. All systemically administered anti-CMV drugs are given in a similar fashion consisting of initial 2-week high-dose treatment (induction) to control the infection followed by long-term lower dose treatment (maintenance) to prevent relapse. Cidofovir is administered as an intravenous infusion once weekly for induction therapy and once every 2 weeks as maintenance therapy. The HPCRT evaluated the efficacy and safety of cidofovir therapy.

The HPCRT was a multicenter, randomized, controlled clinical trial of cidofovir for the treatment of CMV (cytomegalovirus) retinitis. Patients with small peripheral CMV (cytomegalovirus) retinitis lesions (i.e., not at risk of immediate loss of visual acuity) were randomized to immediate treatment with cidofovir or deferred therapy until the retinitis had progressed. Patients randomized to immediate therapy received either 1) low-dose cidofovir at 5 mg/kg once weekly induction for 2 weeks, followed by 3 mg/kg once every 2 weeks for maintenance or 2) high-dose cidofovir at 5 mg/kg once weekly induction for 2 weeks followed by 5 mg/kg once every 2 weeks for maintenance. Patients whose retinitis progressed were given treatment according to best medical judgement, and those assigned to deferral were generally treated with cidofovir.

Outcomes in this trial included retinitis progression, loss of retinal area, and morbidity.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of AIDS according to the Centers for Disease Control and Prevention (CDC)
* 13 years or older
* Diagnosis of CMV (cytomegalovirus) retinitis as determined by a SOCA-certified Ophthalmologist.
* At least one lesion whose size is one-quarter disc area or more that can be photographed.
* Visual acuity in an affected eye of 3 or more lines on the (ETDRS) Early Treatment Diabetic Retinopathy Study chart at 1 meter distance (Snellen equivalent 8/200).
* score of 60 or more on the Karnofsky scale.
* Serum creatinine of 1.5mg/dL or less
* less than 1+ proteinuria on urinalysis
* Total bilirubin of 3.0 mg/dL or less
* Hepatic transaminase levels that do not exceed 5 times the normal levels
* Absolute neutrophil count of 750 cells/µL or greater
* Platelet count of 50,000 cells/µL or greater
* Hemoglobin of 7.5 g/dL or greater
* Negative pregnancy test (females of childbearing potential)
* All men/women of childbearing potential should practice birth control to prevent pregnancy while on study and for 3 months afterwards
* Willingness/ability, with the assistance of a caregiver if necessary to comply with treatment and follow-up procedures
* Signed consent statement

Exclusion criteria:

* Evidence of a CMV (cytomegalovirus) retinitis lesion within zone 1. A lesion less than 1,500 µ from the margin of the optic disc or less than 3,000 µ from the center of the fovea in either eye excludes a patient.
* Evidence of a CMV retinitis lesions that involves 25% or more of the retinal area regardless of location.
* Previous or ongoing therapy for CMV (cytomegalovirus) disease with ganciclovir, foscarnet, CMV hyperimmune immunoglobulin, or other investigational agents solely as prophylaxis are eligible for enrollment.
* Retinal detachment(s) in the affected eye(s)
* media opacity that precludes visualization of the fundus of both eyes.
* patients with a diagnosis of extraocular CMV (cytomegalovirus) disease.
* Patients with history of clinically significant renal disease or renal dialysis.
* Patients with history of clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* pregnant or lactating
* patients with active medical problems including drug or alcohol abuse which could hinder compliance with treatment or follow-up procedures.
* patients receiving therapy within the previous 7 days with nephrotoxic drugs, including: Amphotericin B, Vidarabine, Aminoglycoside antibiotics, Intravenous pentamidine. Patients receiving any of these drugs must discontinue the drug(s) at least one week prior to the time of enrollment, and for the duration of the trial period.
* history of clinically significant probenecid allergy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1994-04; Primary Completion 1996-02 (Actual); Study Completion 1996-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Jabs, MD, Study Chair — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Background] Parenteral cidofovir for cytomegalovirus retinitis in patients with AIDS: the HPMPC peripheral cytomegalovirus retinitis trial. A randomized, controlled trial. Studies of Ocular complications of AIDS Research Group in Collaboration with the AIDS Clinical Trials Group. Ann Intern Med. 1997 Feb 15;126(4):264-74. doi: 10.7326/0003-4819-126-4-199702150-00002. PMID 9036798
- [Background] Long-term follow-up of patients with AIDS treated with parenteral cidofovir for cytomegalovirus retinitis: the HPMPC Peripheral Cytomegalovirus Retinitis Trial. The Studies of Ocular Complications of AIDS Research Group in collaboration with the AIDS Clinical Trials Group. AIDS. 2000 Jul 28;14(11):1571-81. PMID 10983644
- [Background] Kravcik S. Cidofovir for cytomegalovirus retinitis. Ann Intern Med. 1997 Sep 15;127(6):490-1. doi: 10.7326/0003-4819-127-6-199709150-00015. No abstract available. PMID 9313009
- [Derived] Holland GN, Van Natta ML, Goldenberg DT, Ritts R Jr, Danis RP, Jabs DA; Studies of Ocular Complications of AIDS Research Group. Relationship Between Opacity of Cytomegalovirus Retinitis Lesion Borders and Severity of Immunodeficiency Among People With AIDS. Invest Ophthalmol Vis Sci. 2019 May 1;60(6):1853-1862. doi: 10.1167/iovs.18-26517. PMID 31042791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April 1994
Groups:
- Treatment Deferral: IV (in the vein) treatment deferred until retinitis progressed, either:
  5 mg/kg IV (in the vein) of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks, or
  5mg/kg IV (in the vein) once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
  Cidofovir: Three groups:
  1. the deferral group, treatment deferred until retinitis progressed
  2. Low-dose cidofovir group, 5 mg/kg of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks.
  3. High-dose cidofovir group, 5mg/kg once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
- Cidofovir (Low Dose): 5 mg/kg IV (in the vein) of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks
  Cidofovir: Three groups:
  1. the deferral group, treatment deferred until retinitis progressed
  2. Low-dose cidofovir group, 5 mg/kg of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks.
  3. High-dose cidofovir group, 5mg/kg once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
- Cidofovir (High Dose): 5mg/kg IV (in the vein) once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
  Cidofovir: Three groups:
  1. the deferral group, treatment deferred until retinitis progressed
  2. Low-dose cidofovir group, 5 mg/kg of body weight once weekly for two weeks, then maintenance therapy with cidofovir, 3mg/kg once every 2 weeks.
  3. High-dose cidofovir group, 5mg/kg once weekly for 2 weeks, then maintenance therapy with cidofovir, 5mg/kg once every two weeks.
Period: Overall Study
Arm/Group | Treatment Deferral | Cidofovir (Low Dose) | Cidofovir (High Dose)
Started | 26 | 26 | 12
Completed | 26 | 26 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Deferral | Cidofovir (Low Dose) | Cidofovir (High Dose) | Total
Number analyzed (Participants) | 26 | 26 | 12 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 12 | 64
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 24 | 24 | 11 | 59

OUTCOME MEASURES:

1. Primary Outcome: Survival
Time Frame: All patients enrolled will be followed until a common study closing date
Measure: Number; unit: participants
Arm/Group | Treatment Deferral | Cidofovir (Low Dose) | Cidofovir (High Dose)
Number analyzed (Participants) | 26 | 26 | 12
participants
  mortality | 6 | 7 | 3
  progression | 20 | 17 | 5
  va loss of 15 letters | 4 | 6 | 2

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Arm/Group | Treatment Deferral | Cidofovir (Low Dose) | Cidofovir (High Dose)
Serious Adverse Events (participants affected / at risk) | 3/26 | 13/26 | 8/12
Other Adverse Events (participants affected / at risk) | 0/26 | 2/26 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Deferral (N=26) | Cidofovir (Low Dose) (N=26) | Cidofovir (High Dose) (N=12)
Proteinuria 2+ (Blood and lymphatic system disorders) | 3 (4) | 13 (21) | 8 (25)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Deferral (N=26) | Cidofovir (Low Dose) (N=26) | Cidofovir (High Dose) (N=12)
Serum creatinine level >= 133 umol/L (1.5 mg/dL) (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less